CLINICAL TRIAL: NCT06380517
Title: A Randomized Trial of Dichoptic Treatment for Amblyopia in Children 4 to 7 Years of Age
Brief Title: Dichoptic Treatment for Amblyopia in Children 4 to 7 Years of Age
Acronym: ATS23
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); Pediatric Eye Disease Investigator Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATS23; 2UG1EY011751 (NIH)
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Amblyopia
Keywords: Dichoptic; Luminopia; Patching; movie
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Luminopia Group (Experimental): watching dichoptic movies/shows wearing the Luminopia headset prescribed 1 hour per day (treatment time can be split into shorter sessions totaling 1 hour each day) 6 days a week with optical correction, if needed.
  Interventions: Device: Luminopia
- Patching Group (Active Comparator): patching of the fellow eye 2 hours per day (treatment time can be split into shorter sessions totaling 2 hours each day) 7 days per week with optical correction, if needed.
  Interventions: Other: Eye Patch

INTERVENTIONS:
Device: Luminopia — dichoptic movies/shows shown through a virtual reality headset
  Arms: Luminopia Group
Other: Eye Patch — Procedure in which the eye is covered utilizing a patch to increase the strength of the uncovered eye
  Arms: Patching Group

SUMMARY:
In children 4 to 7 years of age, to determine if treatment with 1 hour per day 6 days per week of watching dichoptic movies/shows wearing the Luminopia headset is non-inferior to treatment with 2 hours of patching per day 7 days per week with respect to change in amblyopic eye distance VA from randomization to 26 weeks.

DETAILED DESCRIPTION:
Participants eligible for the study will be randomly allocated (1:1) to receive either dichoptic treatment while wearing the Luminopia headset or patching treatment of the fellow eye for amblyopia with clinical assessments at 13, and 26-weeks post-randomization.

At the 26-week primary outcome visit, participants who were randomly assigned to receive patching treatment with an IOD of 1 logMAR line or more, will be offered Luminopia dichoptic therapy and if they accept, followed forward with visits at 39- and 52-weeks post-randomization.

The study will end for all other participants.

ELIGIBILITY:
At the time of enrollment, individuals must meet all the following inclusion criteria to be eligible to participate in the study.

1. Age 4 to 7 years.
2. Visual acuity, measured in each eye without cycloplegia in current refractive correction (if applicable) using the ATS-HOTV VA protocol on a study-approved device displaying single surrounded optotypes, as follows:

   1. VA in the amblyopic eye 20/40 to 20/200 inclusive.
   2. Age-normal VA in the fellow eye:44,45

      • 4 years: 20/40 or better; 5-6 years: 20/32 or better; 7 years: 20/25 or better
   3. Interocular difference ≥ 3 logMAR lines (i.e., amblyopic eye VA at least 3 logMAR lines worse than fellow eye VA).
3. Amblyopia associated with strabismus, anisometropia, or both (previously treated or untreated).

   1. Criteria for strabismic amblyopia: At least one of the following must be met:

      * Presence of a heterotropia on examination at distance or near fixation (with optical correction), must be <=5 prism diopters (∆) by SPCT at distance and near fixation (see #7 below).
      * Documented history of strabismus which is no longer present (which in the judgment of the investigator could have caused amblyopia).
   2. Criteria for anisometropia: At least one of the following criteria must be met:

      * ≥1.00 D difference between eyes in spherical equivalent (SE).
      * ≥1.50 D difference in astigmatism between corresponding meridians in the two eyes.
   3. Criteria for combined-mechanism: Both of the following criteria must be met:

      * A criterion for strabismus is met (see above).
      * ≥1.00 D difference between eyes in spherical equivalent OR ≥1.50 D difference in astigmatism between corresponding meridians in the two eyes.
4. No more than 2 weeks (cumulative) of prior dichoptic treatment.
5. No treatment with cycloplegic eyedrops (e.g., atropine) in the past 2 weeks; other treatments allowed up to enrollment but then must be discontinued.
6. Refractive correction is required (single vision lenses or contact lenses) for any of the following refractive errors based on a cycloplegic refraction completed within the last 7 months:

   * Hypermetropia of 2.50 D or more by SE
   * Myopia of amblyopic eye of 0.50D or more SE
   * Astigmatism of 1.00D or more
   * Anisometropia of more than 0.50D SE

   NOTE: Monocular or binocular contact lens wear is allowed provided the contact lenses meet the refractive error correction requirements below. For each child, all testing must be performed using the same form of optical correction (i.e., no changing between contacts and spectacles).
   1. Spectacles/contact lens correction prescribing instructions referenced to the cycloplegic refraction completed within the last 7 months:

      * SE must be within 0.50D of fully correcting the anisometropia (if new glasses are prescribed, reduction in plus sphere must be symmetric in the two eyes).
      * SE must not be under corrected by more than 1.50D SE.
      * Cylinder power in both eyes must be within 0.50D of fully correcting the astigmatism.
      * Axis must be within +/- 10 degrees if cylinder power is ≤1.00D, and within +/- 5 degrees if cylinder power is >1.00D.
      * Myopia must not be under corrected by more than 0.25D or over corrected by more than 0.50D SE, and any change must be symmetrical in the two eyes.
   2. Spectacles/contact lens correction (with or without other treatment such as patching) meeting the above criteria must be worn:

      * For at least 18 weeks OR until VA stability is documented (defined as <0.1 logMAR change by the same testing method measured on 2 consecutive exams at least 9 weeks apart).
      * For determining VA stability (non-improvement):

        * The first of two measurements may be made 1) in current correction, or 2) in trial frames with or without cycloplegia or 3) without correction (if new correction is prescribed),
        * The second measurement must be made without cycloplegia in the correct spectacles/contact lens correction that has been worn for at least 9 weeks.
        * NOTE: Because this determination is a pre-randomization, the method of measuring VA is not mandated.
7. Participant is willing to wear the Luminopia headset.
8. Participant is willing to continue full-time spectacles/contact lens wear (if needed).
9. Participant is willing to accept assignment to either dichoptic shows (view 1 hour per day 6 days per week) OR part-time patching (2 hours per day 7 days per week) for 26 weeks.
10. Interpupillary distance of 52mm to 72mm inclusive.
11. Investigator is willing to prescribe Luminopia or patching per protocol.
12. Parent understands the protocol and is willing to accept randomization.
13. Parent has phone (or access to phone) and is willing to be contacted by JAEB Center.
14. Relocation outside area of active PEDIG site within the next 52 weeks is not anticipated.

Individuals meeting any of the following criteria will be excluded from study participation.

1. Heterotropia more than 5∆ at distance or near (measured by SPCT in current correction)
2. Prism lenses or need of a prism prescription at enrollment.
3. Current bifocal spectacles (eligible only if bifocal discontinued 2 weeks prior to enrollment).
4. Myopia greater than -6.00D spherical equivalent in either eye.
5. Previous intraocular or refractive surgery.
6. Known skin reactions to patch or bandage adhesives.
7. Ocular co-morbidity that may reduce VA determined by an ocular examination performed within the past 7 months (Note: nystagmus per se does not exclude the participant if the above visual acuity criteria are met using patch occlusion. Fogging is not permitted).
8. Diplopia more than once per week over the last week prior to enrollment by parental report.
9. History of light-induced seizures.
10. Severe developmental delay that would interfere with treatment or evaluation (in the opinion of the investigator). Participants with mild speech delay or reading and/or learning disabilities are not excluded.
11. Participation in a prior study involving patching for amblyopia
12. Immediate family member (biological or legal guardian, child, sibling, parent) of investigative site personnel directly affiliated with this study or an employee of the JAEB center for Health Research.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 238 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in amblyopic eye logMAR distance VA between randomization and 26 weeks | 26 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Raghuram, OD, PhD, Study Chair — Boston Children's Hospital/ Harvard Medical School; Kammi Gunton, MD, Study Chair — Wills Eye Hospital; Robert Henderson, MS, Principal Investigator — Jaeb Center for Health Research
Locations (72):
- United States (72):
  - UAB Pediatric Eye Care; Birmingham Health Care, Birmingham, Alabama
  - Midwestern University Eye Institute, Glendale, Arizona
  - Phoenix Children's Medical Group - Ophthalmology, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - Arkansas Childrens, Little Rock, Arkansas
  - McFarland Eye Care Center, Little Rock, Arkansas
  - Univ. of California- Berkeley, Berkeley, California
  - Southern California College of Optometry, Fullerton, California
  - Univ of California, Irvine- Gavin Herbert Eye Institute, Irvine, California
  - Children's Hospital of Los Angeles (CHLA), Los Angeles, California
  - Jules Stein Eye Institute at the University of California, Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Western University College of Optometry, Pomona, California
  - University of California, Davis, Sacramento, California
  - Rady Children's Hospital - San Diego Dept of Ophthalmology, San Diego, California
  - University of California San Francisco Department of Ophthalmology, San Francisco, California
  - Yale University, New Haven, Connecticut
  - University of South Florida (USF) Eye, Tampa, Florida
  - The Emory Eye Center, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Illinois College of Optometry, Chicago, Illinois
  - Midwestern University Eye Institute, Downers Grove, Illinois
  - Progressive Eye Care, Lisle, Illinois
  - Indiana School of Optometry, Bloomington, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Dept of Ophthalmology, Prairie Village, Kansas
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Wilmer Eye Institute, Baltimore, Maryland
  - Specialized Pediatric Eye Care, Beverly, Massachusetts
  - New England College of Optometry, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Boston Children's Hospital Waltham, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan College of Optometry at Ferris State Univ, Big Rapids, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Pediatric Ophthalmology, P.C., Grand Rapids, Michigan
  - Children's Eye Care PC, West Bloomfield, Michigan
  - Zenith Vision Development Center, Duluth, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Department of Ophthalmology, Rochester, Minnesota
  - PineCone Vision Center, Sartell, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Ross Eye Institute, University of Buffalo, Med School Dept Ophthalmology, Buffalo, New York
  - NYU Langone Health, New York, New York
  - State University of New York, College of Optometry, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Eye Center, Durham, North Carolina
  - University of North Dakota, Grand Forks, North Dakota
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cole Eye Institute, Cleveland, Ohio
  - Pediatric Ophthalmology Associates, Inc., Columbus, Ohio
  - Ohio State University College of Optometry, Columbus, Ohio
  - Rainbow Babies and Children's Hospital Dept of Ophth, Mayfield Heights, Ohio
  - Eye Care Associates, Inc., Poland, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Pediatric Ophthalmology of Erie, Erie, Pennsylvania
  - Conestoga Eye, Lancaster, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Pennsylvania College of Optometry, Salus at Drexel University, Philadelphia, Pennsylvania
  - Prisma Health, Columbia, South Carolina
  - Storm Eye Institute, Mt. Pleasant, South Carolina
  - Southern College of Optometry, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Children's Hospital - Dept. Of Ophthalmology, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of the Incarnate Word, San Antonio, Texas
  - Earl R. Crouch, III, Norfolk, Virginia
  - Virginia Pediatric Eye Center, Norfolk, Virginia
  - Seattle Children's Hospital, University of Washington, Seattle, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
  - Gundersen Health System, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the Pediatric Eye Disease Investigator Group (PEDIG) public website after the completion of each protocol and publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after publication.
Access Criteria: Users accessing the data must enter an email address.
URL: http://pedig.jaeb.org

DOCUMENTS (3):
  • Study Protocol (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT06380517/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT06380517/SAP_001.pdf
  • Informed Consent Form (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT06380517/ICF_002.pdf